CLINICAL TRIAL: NCT00344045
Title: A Phase IV, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Analgesic Efficacy And Safety of IV Paracetamol Versus Placebo in Subjects With Postoperative Pain After Total Hip Arthroplasty
Brief Title: Study to Evaluate The Analgesic Efficacy and Safety of Intravenous Paracetamol in Subjects With Postoperative Pain After Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN145-010
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: Subjects with postoperative pain after Total Hip Arthroplasty
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Paracetamol
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — IV Solution, Intravenous, 100 mL (10 mg/mL), 4 times at 6-hour intervals, 24 hours
  Other Names: Perfalgan
  Arms: A
Drug: Placebo — IV Solution, Intravenous, 100 mL (0 mg/mL), 4 times at 6-hour intervals, 24 hours
  Arms: B

SUMMARY:
The main purpose is to evaluate the analgesic efficacy of 1g of intravenous (Iv) paracetamol versus i.v. placebo, administered every 6h, as measured by the reduction of the 24-hour cumulative dose of the opioid tramadol in the treatment of postoperative pain following total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Spinal anesth
* BMI 10-35
* No pain conditions/concom med may alter pain quantif.

Exclusion Criteria:

* Other add. surgery
* Liver/Renal function altered
* coagulation alterations
* Respir / Cardiac insufficiency
* Agents affecting microsomal syst

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
24-hour cumulative dose of tramadol | 24 hours, defining TO as the start time of the first dose of study drug

SECONDARY OUTCOMES:
Sum of tramadol and Boluses number, Time from study drug start to tramadol start, total opioid use, Pain intensity scores/diff. from baseline, Global efficacy evaluation, Number of AE, Sedation level, Nausea/Vomiting, Antiemetic needs. | 24 hours, defining TO as the start time of the first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Spain (4):
  - Local Institution, Alcorcón
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Vizcaya